CLINICAL TRIAL: NCT04085211
Title: A Series of Prospective Observational Studies Investigating the Clinical Utility of Image-enhanced Endoscopy in the Gastrointestinal (GI) Tract
Brief Title: Image-Enhanced Endoscopy in the Gastrointestinal Tract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH19-069
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Gastro-Intestinal Disorder; Inflammatory Bowel Diseases; Gastro Esophageal Reflux; Atrophic Gastritis; Neuroendocrine Tumors
Keywords: endoscopy
MeSH Terms: conditions — Digestive System Diseases; Inflammatory Bowel Diseases; Gastroesophageal Reflux; Gastritis, Atrophic; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Inflammatory Bowel Disease: Patients with an established diagnosis of ulcerative colitis or Crohn's Disease who require either a flexible sigmoidoscopy or colonoscopy as part of routine care (e.g. surveillance or staging disease activity)
- Patients with symptoms of gastro-oesophageal reflux disease: Patients with symptoms of gastro-oesophageal reflux disease requiring a gastroscopy as part of routine clinical care.
- Atrophic gastritis: Patients with known or suspected atrophic gastritis that require a gastroscopy to either confirm the diagnosis or surveillance for pre-cancerous changes.
- Neuroendocrine Tumours: Patients with an established history of gastric neuroendocrine tumours requiring surveillance

SUMMARY:
This study evaluates a range of endoscopic image enhancement techniques for assessing conditions involving the gastrointestinal tract.

This study aims to determine:

(i) the accuracy of different techniques to diagnose or grade severity of several gastrointestinal conditions

(ii) if image-enhancement techniques could potentially replace investigations currently used in daily practice (e.g. biopsy) with a view to reduce costs and shorten the interval to initiate treatment

DETAILED DESCRIPTION:
Endoscopic procedures are performed on a daily basis to visualise the gastrointestinal tract for diagnosis and intervention. The demand for procedures is growing, consequently increasing the number of additional investigations; for example, biopsies. Image enhancement techniques can be performed during procedures either digitally or through the use of dye. These techniques alter the qualities of the image e.g. colour, contrast and magnification. We believe these techniques have several potential benefits: (i) improve diagnostic accuracy (ii) filter appropriate selection of additional investigations to maximise diagnostic yield (iii) the potential to replace existing investigations which are costly and intricate.

Participants included in the study will have an endoscopic procedure as indicated for routine clinical care. On the day of the procedure (or before), a baseline assessment will be performed - symptom questionnaires, medical history and recording any relevant investigation results performed as part of routine care. Participants will have the endoscopic procedure as normal, with additional images and video obtained using different image enhancement techniques. Select patients will have follow-up for up to one year to determine relapse. The image enhancement technique findings will be compared to the gold standard investigation currently available as part of routine care for the condition of interest.

The study will look at a range of different image enhancement techniques: dye chromoendoscopy, blue laser imaging (BLI), linked colour imaging (LCI), narrow band imaging (NBI), image magnification and endocytoscopy. This will involve a range of gastrointestinal conditions.

Ethics Approval: favourable opinion was provided by the East Midlands - Derby research and ethics committee, reference: 19/EM/0167.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patient has mental capacity to consent
* Requires endoscopic procedure as part of routine care

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from a hospital setting, predominantly an outpatient setting where an endoscopic procedure is required part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value of specific endoscopic image enhancement findings to diagnose or stage the severity of different gastrointestinal conditions | 8 weeks
  Identify specific features on NBI,BLI, LCI, magnification and endocytoscopy to accurately diagnose / grade severity of a range of conditions when compared to the gold standard diagnostic investigation e.g. biopsy, pH impedance testing

SECONDARY OUTCOMES:
Specific image enhancement findings to predict relapse for patients with inactive inflammatory bowel disease. | 12 months
  Relapse as defined by the requirement for treatment escalation, surgery, hospital admission; biochemical evidence of relapse (faecal calprotectin) or worsening inflammation on repeat endoscopy.
median duration for image enhanced endoscopy procedures | 1 day
  median duration (minutes) as defined as the time interval between insertion and completed withdrawal of the endoscope

CONTACTS AND LOCATIONS:
Overall Officials: Bu'Hussain Hayee, PhD, MBBS,, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- Department of Gastroenterology, King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided